CLINICAL TRIAL: NCT04300608
Title: Functional and Metabolomic Biomarkers of Mitochondrial Dysfunction in Parkinson's Disease
Brief Title: Measures of Mitochondria Dysfunction in PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, David Marcinek, Professor of Radiology Research, University of Washington
Other Study IDs: STUDY00007024
Record Dates: First submitted 2020-03-03; First posted 2020-03-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease, Mitochondrial
Keywords: Parkinson Disease; Mitochondria; Skeletal Muscle; Bioenergetics
MeSH Terms: conditions — Parkinson Disease, Mitochondrial; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates metabolic and functional parameters in the skeletal muscle of Parkinson's disease patients for comparison to a set of healthy age-matched controls.

DETAILED DESCRIPTION:
The goal of this study is to identify the unique signature of bioenergetic markers and mitochondrial (dys)function in muscle of individuals with PD, who are 65-85 of age, read and speak English, have a Hoehn & Yahr score between 2 and 3 (bilateral disease, not severely disabled) and have a clinical diagnosis of PD. Bioenergetic markers and muscle functional properties will be compared to a control dataset collected over the last few years from healthy elderly subjects in the same age range to provide a foundation for future intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85 years.
* Ability to attend a 3-hour study visit in Seattle, WA.
* Ability to read and speak English.
* Hoehn & Yahr Stage 2-3. (bilateral disease, not severely disabled.)

Exclusion Criteria:

* Any contra-indication to magnetic resonance imaging
* A history of epilepsy, stroke, brain surgery, or structural brain disease.
* The presence of other serious illnesses
* Current or recent enrollment in a clinical trial involving an investigational product or device.
* Supplementation with NAD, nicotinamide mononucleotide (NMN), nicotinamide riboside (NR), and other nutraceuticals designed to target NAD for 30 days prior to baseline study visit.
* Current drug or alcohol use or dependence.
* Inability/unwillingness to provide informed consent. (e.g. diagnosis of dementia, confusion about study goals or participation.)
* Acute infection (e.g. upper respiratory, dermal) in the previous 30 days.
* Right limb tremor or dyskinesia that cannot be comfortably controlled for 90 minutes.

Ages: 65 Years to 85 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients diagnosed with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
ATPmax | baseline
  Maximal mitochondrial ATP production rates measured by magnetic resonance spectroscopy
NAD(H) metabolites | baseline
  Measurement of relative NAD(H) metabolite concentrations in resting skeletal muscle by magnetic resonance spectroscopy
Muscle force and endurance | baseline
  Maximum voluntary contraction (MVC) force in Newtons and fatigue resistance assessed by the ability to maintain repeated contractions at 70% MVC will be measured in the hand (flexor digitorum interroseus) and leg (tibialis anterior) using isometric contractions in a custom made apparatus.

SECONDARY OUTCOMES:
Mitochondrial metabolites | baseline
  Separate measurement of NAD(H) metabolite concentrations in cytosol and mitochondria by magnetic resonance spectroscopy in resting skeletal muscle
Relationship between self report function and mitochondrial energetics | baseline
  Correlation between self report of fatigue, balance, and muscle pain (PRO-PD) with ATPmax rates and NAD(H) metabolite concentrations measured using magnetic resonance spectroscopy.
Relationship between clinical assessment and mitochondrial energetics | baseline
  Correlation between UPDRS with ATPmax and NAD(H) metabolites

CONTACTS AND LOCATIONS:
Overall Officials: David Marcinek, PhD, Principal Investigator — University of Washington; Laurie Mischley, ND, MPH, PhD, Principal Investigator — Bastyr University
Locations (1):
- University of Washington, Seattle, Washington, United States